CLINICAL TRIAL: NCT03596047
Title: Clinical Trial With Random Assignment to Evaluate the Efficacy and Safety of Radial Waves for the Treatment of Erectile Dysfunction
Brief Title: Radial Shockwave Therapy for Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMGC-4
Record Dates: First submitted 2018-06-13; First posted 2018-07-23 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
Keywords: radial wave therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Shockwave therapy machine has a device to prevent the patient from receiving the radial wave. This device will be changed for the clinic administrator.
  Change device placebo wave therapy, using the respective device t
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment + Radial wave therapy (Experimental): Sildenafil according to the degree of patient involvement + 6 sessions of radial waves.
  Interventions: Device: Radial wave therapy
- Standard treatment + Placebo therapy (Placebo Comparator): Sildenafil according to the patient's degree of affectation + 6 sessions of placebo therapy.
  Interventions: Device: Placebo therapy

INTERVENTIONS:
Device: Radial wave therapy — 6 radial waves' sessions. A weekly session of radio waves will be applied with the following parameters: 6000 pulses at 1.5-2.6 bar (depending on patient tolerance), with a frequency of 12Hz, the frequency should increase to 17HZ the first 500 impulses to create mild anesthesia in the area; in all the sessions of radial waves, 4000 impulses will be distributed in the body of the penis in scanning technique and 2000 impulses in the perineal area, specifically in the ischiocavernosus and bilateral bulbo-sponge muscles. During the period of therapy application, patients will receive oral treatment with sildenafil according to the patient's degree of affectation.
  Arms: Standard treatment + Radial wave therapy
Device: Placebo therapy — There will be a weekly session of placebo wave therapy, using the respective device to prevent the patient from receiving the radial wave. The same parameters of the "real" therapy will be used: 6000 pulses at 2.6 bar, with a frequency of 17 Hz; in all the sessions of radial waves, 4000 impulses will be distributed in the body of the penis in scanning technique and 2000 impulses in the perineal area. During the period of therapy application, patients will receive oral treatment with sildenafil according to the patient's degree of affectation.
  Arms: Standard treatment + Placebo therapy

SUMMARY:
Objective: To evaluate the efficacy and safety of radial shock waves for the treatment of erectile dysfunction [ED].

Patients and methods: Randomized, double-blind clinical trial. The study will include patients of legal age with diagnosis of ED and score on the International Index of Erectile Function [IIEF-EF] scale between 11 and 21 points, who voluntarily decide to participate and sign the informed consent. Patients with bladder cancer, prostate cancer or active colon, ED of psychological origin, any psychiatric disorder, spinal cord injury, clinical suspicion of hypogonadism (score on the Aging Males' Symptoms scale greater than 36), infections or active lesions of the penis or pubic area, ED secondary to treatment with medications (antiandrogenic therapy, use of corticosteroids, anti-Parkinson's, antipsychotics), radical prostatectomy or other radical pelvic surgery, history of pelvic radiotherapy, penile implantation, or endocrine diseases that occur with ED (acromegaly, gigantism, Addison's disease, hyperprolactinemia, androgenic deficiency), sickle cell anemia, and anticoagulated patients will be excluded.

Patients will be randomly assigned to one of the following treatment arms:

* Arm 1 (Standard treatment (oral sildenafil) + Radial wave therapy)
* Arm 2 (Standard treatment (oral sildenafil) + Placebo therapy)

Measurements will be made of the Erection Hardness Score [EHS] and IIEF-EF scale scores, of the use of medication and of the possible adverse events of the therapy, at the beginning and end of the treatment, and one month after the therapies are finished.

DETAILED DESCRIPTION:
Background: Radial shock waves are an effective therapy for the management of various problems at the muscular and joint level, thanks to the effect it has on the activation of microcirculation. The effect of these waves on patients with erectile dysfunction is currently unknown; however, it is considered possible to help recovery in patients with vascular origin dysfunction by increasing microcirculation blood flow in this area.

Objective: To evaluate the efficacy and safety of radial shock waves for the treatment of erectile dysfunction.

Patients and methods: Randomized, double-blind clinical trial. The study will include patients of legal age with diagnosis of ED and score on the IIEF-EF scale between 11 and 21 points, who voluntarily decide to participate and sign the informed consent. Patients with bladder cancer, prostate cancer or active colon, ED of psychological origin, any psychiatric disorder, spinal cord injury, clinical suspicion of hypogonadism (AMS greater than 36), infections or active lesions of the penis or pubic area, ED secondary to treatment with medications (antiandrogenic therapy, use of corticosteroids, anti-Parkinson's, antipsychotics), radical prostatectomy or other radical pelvic surgery, history of pelvic radiotherapy, penile implantation, or endocrine diseases that occur with ED (acromegaly, gigantism, Addison's disease, hyperprolactinemia, androgenic deficiency), sickle cell anemia, and anticoagulated patients will be excluded.

Patients will be randomly assigned to one of the following treatment arms:

* Arm 1 (Standard treatment (oral sildenafil) + Radial wave therapy): Sildenafil according to the degree of patient involvement + 6 sessions of radial waves. A weekly session of radial waves will be applied with the following parameters: 6000 pulses at 1.5-2.6 bar (depending on patient tolerance), with a frequency of 17Hz, the frequency should increase to 22HZ the first 500 impulses to create mild anesthesia in the area; in all radial wave sessions, 4000 impulses will be distributed in the body of the penis in scanning technique and 2000 impulses in the perineal area.
* Arm 2 (Standard treatment (oral sildenafil) + Placebo therapy): Sildenafil according to the patient's degree of affectation + 6 sessions of placebo therapy. There will be a weekly session of placebo wave therapy, using the respective device to prevent the patient from receiving the radial wave. The same parameters of the "real" therapy will be used: 6000 pulses at 2.6 bar, with a frequency of 17 Hz; in all radial wave sessions, 4000 impulses will be distributed in the body of the penis in scanning technique and 2000 impulses in the perineal area.

Measurements will be made of the EHS and IIEF-EF scale scores, of the use of medication and of the possible adverse events of the therapy, at the beginning and end of the treatment, and one month after the therapies are finished.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 18 years
* Erectile dysfunction present more for more than 3 months in more than 50% of intercourse.
* IIEF-EF score between 11 and 21.
* Patient who agrees to enter the study through the signing of an informed consent.

Exclusion Criteria:

* EHS score of 4
* Bladder, prostate or colon cancer.
* ED of psychological origin.
* Patients with spinal cord injury.
* Patients with anticoagulant use.
* Patients with sickle cell anemia.
* Patients with clinical suspicion of hypogonadism (AMS greater than 36, Annex 1).
* Patients with infections or active lesions of the penis or pubic area.
* Patients with ED secondary to drug treatment (antiandrogenic therapy, antidepressants, use of corticosteroids, antiparkinsonians, antipsychotics).
* Radical prostatectomy or other radical pelvic surgery.
* Antecedents of pelvic radiotherapy.
* Patients with penile implant.
* Endocrine diseases that occur with ED: acromegaly, gigantism, Addison's disease, hyperprolactinemia, androgenic deficiency.
* Patients with neurological diseases (Parkinson's, CVD, dementia of any origin)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Saffon, Doctor, Principal Investigator — Boston Medicval Group
Locations (1):
- Boston Medical Group Colombia, Bogotá, Cundinamarca, Colombia

REFERENCES:
- [Derived] Sandoval-Salinas C, Saffon JP, Martinez JM, Corredor HA, Gallego A. Are Radial Pressure Waves Effective for the Treatment of Moderate or Mild to Moderate Erectile Dysfunction? A Randomized Sham Therapy Controlled Clinical Trial. J Sex Med. 2022 May;19(5):738-744. doi: 10.1016/j.jsxm.2022.02.010. Epub 2022 Mar 24. PMID 35341724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out in two clinics over a period of 26 months.
Period: Overall Study
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy
Started | 40 | 40
Completed | 33 | 34
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.8) | 48.5 (11.2) | 48 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.7 (3.7) | 26.8 (3.3) | 26.75 (3.5)
International Index of Erectile Function-Erectile Function domain [Mean (Standard Deviation); unit: units on a scale] — The scale score ranges from 0 to 30, a score less than 26 is considered to have erectile dysfunction. Using the IIEF-EF, erectile dysfunction severity categories are no ED (score ≥26 out of 30) mild (score 22-25), mild-to-moderate (score 17-21), moderate (score 11-16), and severe (score ≤10)
  units on a scale | 16.3 (3.2) | 16.4 (3.2) | 16.3 (3.2)
Erection Hardness Score [Median (Full Range); unit: units on a scale] — The Erection Hardness Score (EHS) is a method to quantify erection outcome data. The score range is from 0 to 4. The EHS is a single-item Likert scale including the following response modalities: 0: "penis does not enlarge," 1: "penis is larger but not hard," 2: "penis is hard but not hard enough for penetration," 3 "penis is hard enough for penetration but not completely hard," and 4 "penis is completely hard and fully rigid"
  units on a scale | 3 [1 to 3] | 3 [2 to 3] | 3 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Change IIEF-EF Score
Description: The scale IIEF-EF score ranges from 0 to 30, a score less than 26 is considered to have erectile dysfunction. Using the IIEF-EF, erectile dysfunction severity categories are no ED (score ≥26 out of 30) mild (score 22-25), mild-to-moderate (score 17-21), moderate (score 11-16), and severe (score ≤10). The difference in the average score of the International Index Erectile Function-Erectile Function domain (IIEF-EF) scale in at least 5 points, between the score at the end of the treatment (6 weeks) and the basal score.
Time Frame: 6 weeks (The end of the treatment)
Population: Patients with results at the end of therapy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy
Number analyzed (Participants) | 33 | 36
units on a scale | 3.4 [1.6 to 5.3] | 4.2 [2.5 to 5.9]

2. Secondary Outcome: IIEF-EF Score After One Month of Follow-up
Description: as for outcome 1
Time Frame: Month 1 of follow-up (Week 10)
Population: Patients with results at week 10
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy
Number analyzed (Participants) | 33 | 34
units on a scale | 0.72 [-1.4 to 2.8] | 2.3 [0.26 to 4.1]

3. Secondary Outcome: Erection Hardness Score (EHS)
Description: Erection Hardness Score (EHS), it is a unique Likert scale. EHS is a self-reported tool that scores erection hardness on a 4-point scale: 0, penis does not enlarge; 1, penis is larger but not hard; 2, penis is hard but not hard enough for penetration; 3, penis is hard enough for penetration but not completely hard; 4: penis is completely hard and fully rigid.
  This outcome is the number of patients that increased the EHS by at least 1 point at week 6 after randomization
Time Frame: 6 weeks (At the end of treatment)
Population: Patients with the results at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy
Number analyzed (Participants) | 33 | 34
Participants | 15 | 14

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Treatment + Radial Wave Therapy | Standard Treatment + Placebo Therapy
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39
Other Adverse Events (participants affected / at risk) | 2/37 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment + Radial Wave Therapy (N=37) | Standard Treatment + Placebo Therapy (N=39)
Not serius (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Facial flushing
Not serius (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Superficial abrasions of the dermis in the penis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03596047/Prot_SAP_000.pdf